CLINICAL TRIAL: NCT04317222
Title: Early Postoperative Continuous Renal Replacement Therapy After Liver Transplantation in Acute-on-chronic Liver Failure Patients With Overt Hepatic Encephalopathy
Brief Title: Early Postoperative CRRT After Liver Transplantation in ACLF Patients With Overt HE
Acronym: LTeCRRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Huimin Yi, Principal Investigator and the director of transplant intensive care unit, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTeCRRT-P1
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Acute-On-Chronic Liver Failure; Hepatic Encephalopathy
Keywords: Acute-On-Chronic Liver Failure; Overt Hepatic Encephalopathy; Continuous Replacement Renal Therapy; Liver Transplantation
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hepatic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eCRRT group (Experimental): Initiated CRRT within the first 24 post-transplant hours.
  Interventions: Device: eCRRT
- Control group (No Intervention): Standard treatment.

INTERVENTIONS:
Device: eCRRT — eCRRT was define as:
  1. Initiated within the first 24 post-transplant hours;
  2. High volume (35-50ml/kg) hemofiltration;
  3. Continuous at least 12 hours per day for 3 days;
  4. Standard treatment
  Arms: eCRRT group

SUMMARY:
Pretransplant hepatoencephalopathy (HE) markedly impacts recipient outcomes after liver transplantation. Intraoperative CRRT showed benefits but feasibility was much concerned. This study aims to observe the effect on consciousness recovery when initiating CRRT early in the post-transplant period in recipients with ACLF and overt HE.

DETAILED DESCRIPTION:
Hepatoencephalopathy (HE) is a common severe decompensation in end stage liver diseases and resulted to the need of liver transplantation (LT). Pretransplant HE markedly impacts recipient outcomes after liver transplantation. HE in acute on chronic liver failure (ACLF) is categorized to type C HE. Hyperammonemia and systemic inflammation have been reported to contribute its development. Continuous renal replacement therapy (CRRT) has been shown great benefits in ACLF patients with HE. Intraoperative CRRT in LT also showed benefits but feasibility was much concerned. Our preliminary retrospective data showed that early CRRT (eCRRT) after LT reduced consciousness recovery time, ventilation days and post-transplant infection rate.

This open label, parallel randomized trial will observe the effect on consciousness recovery when initiating CRRT early (eCRRT) in the post-transplant period in recipients with ACLF and overt HE.

The CRRT safety and ventilation days, infection, mortality and ICU stay will also be measured.

ELIGIBILITY:
Inclusion Criteria: Liver transplant recipients who meet all of the following criteria will be enrolled

1. Pre transplant liver failure: Total bilirubin over 171μmol/L and prothrombin activity (PTA)<40%;
2. Overt hepatic encephalopathy(HE): Grade II or higher HE according West Haven classification;
3. HE associated with acute liver failure (Type A) or cirrhosis complicated with portal hypertension and/or portal systemic shunts (Type C)

Exclusion Criteria:

1. Patients with a previous history of kidney-related diseases and glomerular filtration rate <30 millilitre per minute;
2. Patients with acute renal failure need CRRT before transplantation;
3. Patients newly developed acute renal failure need CRRT at the time of randomization;
4. Retransplantation or multiple-organs transplantation;
5. Any ischemic or hemorrhagic stroke co-morbidity;
6. Hemodynamic instability requiring fluid resuscitation or very high dose of vasopressors;
7. Extremely moribund patients with an expected life expectancy of less than 24 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Consciousness recovery time | From the immediate to 30 days after liver transplantation
  The period from post-transplant immediate to the time when the patient have the first spontaneous eye opening and proper motor response to commands.
Adverse events | From the immediate to 7 days after liver transplantation (CRRT therapy period)
  Any adverse event which probable related with CRRT

SECONDARY OUTCOMES:
Invasive ventilation days | From the immediate to 30 days after liver transplantation
  The time period when patients breath with ventilator through artificial airway
ICU stay (days) | up to one year
  The time period from transplantation to first ICU discharge
Reintubation rate | From the immediate to 30 days after liver transplantation
  Reintubation after the first extubation following liver transplantation
90 days mortality | From the immediate to 90 days after liver transplantation
  All cause mortality
Infection rate | From the immediate to 30 days after liver transplantation
  Any diagnosed infection after transplantation in 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Huimin Yi, MD, Principal Investigator — The 3rd affiliated hospital of Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data (IPD) that underlie results in a publication will be shared with other researchers.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: One year from the time of result publication
Access Criteria: Claim from Principle investigator by email. Need Curriculum Vitae.

REFERENCES:
- [Result] Yi H, Lv H, An Y, Yi X, Wei X, Chen G (2015) Early Continuous Blood Purification(CBP) Deceased the Incidence of Pulmonary Infection after Liver Transplantation in Severe End-Stage-Liver-Disease Recipients With Hepatic Encephalopathy. Transplantation 99:201-201